CLINICAL TRIAL: NCT06015321
Title: Open Label Trial of Maintenance Enzalutamide in CRPC
Brief Title: An Open Label Phase II Study of First-Line Maintenance Enzalutamide Following Docetaxel Plus Androgen-Deprivation Therapy in Patients With Previously-Untreated, Metastatic, Castration-Naive Prostatic Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Sung Hee Lim, Samsung Medical Center, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-07-103
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Prostatic Adenocarcinoma
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enzalutamide (Experimental): First-Line Maintenance Enzalutamide Following Docetaxel plus Androgen-Deprivation Therapy in Patients with Previously-Untreated, Metastatic, Castration-Naïve Prostatic Adenocarcinoma
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — enzalutamide 160 mg PO daily
  Other Names: XtandiTM

SUMMARY:
Although surgical or medical castration (i.e., androgen-deprivation therapy, ADT) is considered standard treatment in metastatic castration-naïve PC (mCNPC) patients, current guidelines have established the addition docetaxel or modern androgen receptor targeting agents (ARTAs; abiraterone acetate or enzalutamide) to ADT as the standard of care for patients with mCNPC [1,2]. One of the major challenges in the management of mCNPC includes balancing the toxicity of first-line docetaxel with clinical benefit. Our previous clinical studies suggested that the tolerability of docetaxel could be improved by using a biweekly regimen [3,4], without compromising efficacy. There is a growing interest in maintenance therapy as a strategy for prolonging the benefit of first-line therapy while minimizing long-term toxicity. In phase III trials involving first-line enzalutamide in mCNPC (ENZAMET and ARCHES), earlier treatment with docetaxel was permitted [5,6]. Based on these considerations, we hypothesized that enzalutamide maintenance therapy would improve outcomes in patients who had received first-line biweekly docetaxel plus ADT for mCNPC.

DETAILED DESCRIPTION:
1. Patients will receive docetaxel 40 mg/m2 IV every 2 weeks plus ADT. Docetaxel will be repeated on an outpatient basis and continued until disease progression, unacceptable toxicity, deterioration of clinical condition, patient refusal, or up to 6 to 8 cycles. ADT includes commercially available GNRH agonists such as goserelin, leuprolide and triptorelin, according to their market authorized approved label.
2. After the receipt of 6 to 8 cycles of first-line docetaxel plus ADT, patients with no evidence of disease progression (i.e., biochemical and clinical) will receive enzalutamide 160 mg PO daily. Enzalutamide will be continued until disease progression (i.e., development of mCRPC), unacceptable toxicity, deterioration of clinical condition, patient refusal.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion of a subject in the study, all of the following inclusion criteria must be fulfilled:

  1. Subject is a male at least 20 years of age.
  2. Subject has a histologically or cytologically confirmed diagnosis of adenocarcinoma of prostate.
  3. Subject has radiologic and clinical evidence of metastatic disease initially or after treatment for localized disease. They must have metastatic or progressive disease for which there is no further curative treatment available.
  4. Subject has an ECOG performance status of 0 to 1.
  5. Subject has a life expectancy of 3 months or more.
  6. At least 4 weeks since the last surgical procedures or radiotherapy prior to enrolment. Subjects must have recovered to <Grade 2 from all acute toxicities or toxicity must be deemed irreversible by the investigator.
  7. Acceptable liver function:
  8. Acceptable renal function
  9. Acceptable hematologic status (without growth factor support or transfusion dependency):
  10. Subject must agree to use an adequate method of contraception (condom) if he is having sex with a woman of childbearing potential or with a woman who is pregnant.
  11. Written and voluntary informed consent understood, signed and dated.

Exclusion Criteria:

For inclusion of a subject in the study, any of the following inclusion criteria must not be fulfilled:

1. Ongoing treatment with an anticancer agent not contemplated in this protocol
2. Pathologic finding consistent with neuroendocrine or small cell carcinoma
3. Any history of clinically relevant coronary artery disease or myocardial infarction within the last 3 years, New York Heart Association (NYHA) grade III or greater congestive heart failure, cerebrovascular attack within the prior year, or current serious cardiac arrhythmia requiring medication except atrial fibrillation.
4. Known uncontrolled brain, leptomeningeal or epidural metastases (unless treated and well controlled for at least 4 weeks prior to Cycle 1 Day 1). Subjects that develop brain metastasis during the study may have their treatment interrupted to receive a course of cranial radiation and restart trial medication after a recovery period of at least 1 week. High dose corticosteroids may be employed for the management of cranial radiation but must be tapered off before resuming treatment.
5. Non-tolerable >Grade 2 neuropathy or evidence of unstable neurological symptoms within 4 weeks of Cycle 1 Day 1.
6. Major surgery, other than diagnostic surgery, within 4 weeks prior to Cycle 1 Day 1, without complete recovery.
7. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
8. Subjects who have exhibited allergic reactions to taxanes.
9. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this study.
10. The subject has legal incapacity or limited legal capacity. Dementia or significantly altered mental status that would limit the understanding or rendering of informed consent and compliance with the requirements of this protocol. Unwillingness or inability to comply with the study protocol for any reason.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subject is a male at least 20 years of age
Enrollment: 51 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Time-to-CRPC (biochemical or clinical) | up tp 30months
  RECIST v1.1 criteria will be used to assess patient response to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR